CLINICAL TRIAL: NCT02562703
Title: Transcutaneous Vagus Nerve Stimulation for Treating Major Depressive Disorder: a Phase II, Randomized, Double-blind Clinical Trial
Brief Title: tVNS for Depression
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Santa Casa Medical School (Other)
Responsible Party: Principal Investigator, Pedro Shiozawa, Coordinator - Interdisciplinary Center for Clinical Neuromodulation, Santa Casa Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tVNS
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACTIVE tVNS (Active Comparator): tVNS will be applied by the external simulator (Monarch). The stimulation will be conducted at a frequency of 120 Hz with pulse duration of 250 microseconds. The current intensity will be individually established and should be equivalent to a slight feeling of not painful paresthesia .The stimulus generates a pulse and asymmetric biphasic waveform. Electrodes (25cm2) will be placed over the mastoid process bilaterally. The study protocol will follow the rational of our previous trials with TNS.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation
- SHAM tVNS (Sham Comparator): tVNS will be applied by the external simulator (Monarch). The stimulation will be turned off after 60 seconds following previous trials.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — tVNS will be applied by the external simulator (Monarch). The stimulation will be conducted at a frequency of 120 Hz with pulse duration of 250 microseconds. The current intensity will be individually established and should be equivalent to a slight feeling of not painful paresthesia .The stimulus generates a pulse and asymmetric biphasic waveform. Electrodes (25cm2) will be placed over the mastoid process bilaterally. The study protocol will follow the rational of our previous trials with TNS.

SUMMARY:
This is a phase II, randomized, sham controlled, clinical trial. This clinical trial has as primary objective to evaluate changes in depressive symptoms of a transcutaneous Vagus Nerve Stimulation (tVNS) treatment protocol for patients with moderate / severe depressive episode.

ELIGIBILITY:
Inclusion Criteria:

1. patients between 18 and 69 years
2. patients with a diagnosis of depression according to the SCID
3. score greater than or equal to 18 on the Hamilton Rating Scale 17-item version (equivalent to moderate or severe depressive episode)
4. agreement to participate in the study as recommended in the IC.

Exclusion Criteria:

1. patients with psychiatric indication for hospitalization
2. patients with psychiatric comorbidity
3. patients with a diagnosis of personality disorder
4. presence of severe neurological or medical diseases such as neoplasms in activity, neurodegenerative diseases and chronic diseases uncompensated.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-02 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
• Hamilton Depressive Rating Scale version 17 items (HDRS-17) | Change from baseline in depressive symptoms at 2 weeks
  This clinical trial has as primary objective to evaluate the effect of the tVNS on depressive symptoms measured by the Hamilton Depressive Rating Scale version 17 items (HDRS-17) in patients with moderate / severe depressive episode.

REFERENCES:
- [Result] Trevizol AP, Sato IA, Bonadia B, Liquidato BM, Barros MD, Cordeiro Q, Shiozawa P. Trigeminal Nerve Stimulation (TNS) for Major Depressive Disorder in Pregnancy: A Case Study. Brain Stimul. 2015 Sep-Oct;8(5):988-9. doi: 10.1016/j.brs.2015.07.034. Epub 2015 Jul 23. No abstract available. PMID 26358492
- [Result] Shiozawa P, Duailibi MS, da Silva ME, Cordeiro Q. Trigeminal nerve stimulation (TNS) protocol for treating major depression: an open-label proof-of-concept trial. Epilepsy Behav. 2014 Oct;39:6-9. doi: 10.1016/j.yebeh.2014.07.021. Epub 2014 Aug 23. PMID 25150403
- [Result] Cook IA, Schrader LM, Degiorgio CM, Miller PR, Maremont ER, Leuchter AF. Trigeminal nerve stimulation in major depressive disorder: acute outcomes in an open pilot study. Epilepsy Behav. 2013 Aug;28(2):221-6. doi: 10.1016/j.yebeh.2013.05.008. Epub 2013 Jun 14. PMID 23773978